CLINICAL TRIAL: NCT03419507
Title: Comparison of a Macintosh Laryngoscope and Endotracheal Tube Introducer During Chest Compression in a Manikin: Randomized, Prospective, Cross-over Study
Brief Title: A Comparison of a Macintosh Laryngoscope and Endotracheal Tube Introducer in a Manikin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hüseyin Cahit Halhallı, MD, Derince Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2017/16. 15/351
Record Dates: First submitted 2018-01-18; First posted 2018-02-05 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Difficult Intubation
Keywords: endotracheal tube introducer; manikin; chest compression

STUDY DESIGN:
Intervention Model Description: Equal numbers 1 and 2 will be written on the same sized papers. After separating participants into two groups, doctors that drawed envelop number 1 will be asked to intubate with No. 3 Macintosh laryngoscopy and doctors that drawed envelop number 2 will be asked to intubate with endotracheal tube introducer. Than groups will be changed.
Who Masked: Participant
Masking Description: The doctors will be informed about the research, but they will be blind to the specific purposes of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Macintosh group (Active Comparator): After separating participants into two groups, doctors that drawed envelop number 1 will be asked to intubate with laryngoscope by using No. 3 Macintosh laryngoscope
  Interventions: Device: Macintosh laryngoscopy
- Endotracheal tube introducer group (Active Comparator): After separating participants into two groups, doctors that drawed envelop number 2 will be asked to intubate with laryngoscope by using the adult size endotracheal tube introducer with using No. 3 Macintosh laryngoscope.
  Interventions: Device: Endotracheal tube introducer

INTERVENTIONS:
Device: Endotracheal tube introducer — The doctors that drawed envelop number 2 will be asked to intubate with laryngoscope by the adult size, endotracheal tube introducer with using No. 3 Macintosh blade
  Arms: Endotracheal tube introducer group
Device: Macintosh laryngoscopy — The doctors who drawed envelope number 1 will asked to intubate with using No. 3 Macintosh blade
  Arms: Macintosh group

SUMMARY:
In this prospective, randomized, cross-over study, investigators aimed to compare the first pass successes of inexperienced doctors with Macintosh laryngoscopy and endotracheal tube introducer on a manikin with continuous chest compression in the ambulance simulation in the pre-hospital process.

DETAILED DESCRIPTION:
This study is a prospective, cross-over manikin study which is based on an ambulance simulation. Written inform consent was obtained from all doctors who agreed to participate to the study. Inexperienced doctors who attended in Kocaeli between February 2018 and March 2018 will be included to the survey. Novice doctors participated to this research. The research will be carried out in the department of emergency medicine of Derince training and research hospital. In order to prevent bias, the eight-hour training module for the participants , theoretical and practical airway training will be provided by an emergency medical specialist who has no knowledge about the research.

The participants will be informed about the study after the training. Doctors who participate to the study will be included after the written inform consent is obtained. The participants will be informed about the research, but they will be blind to the specific purposes of the study. The participants will practice for 5 minutes on the manikin by themselves and with the emergency medicine specialist if they ask for. Life / form® Deluxe Crisis ™ Manikin Torso with Advanced Airway Management will be used as the research manikin. The participants will perform airway interventions in the sitting position and the height of the stretcher will be set at the same height with the ambulance stretcher. Practitioner's seat will be set on the same height with the ambulance seat. 8.0 (mm ID) endotracheal tube will be used for the procedure. Endotracheal tube and manikin airway will be lubricated with pump spray lubricant provided with the simulator. Airway manikin will be in supine position. Lund University Cardiac Arrest System-version 2 (LUCAS 2TM) automatic chest compression device will be used to provide 5 cm compression depth and 100 chest compressions per minute in order to provide standardization in chest compression and prevent bias created by practitioners. The airway devices will be next to the model's head.

The study was planned as a randomized, crossover clinical trial to reduce the influence of the learning. Equal numbers 1 and 2 will be written on the same sized papers to provide randomization. All papers will be folded in the same way and placed inside brown and invisible envelopes. All of the envelopes will be placed in the same box. After the training, every doctor will be asked to choose one of the envelopes. After separating the participants into two groups, doctors that drawed envelop number 1 will be asked to intubate by using only No. 3 Macintosh blade. The doctors that drawed envelop number 2 will be asked to intubate with the adult size endotracheal tube introducer with using No. 3 Macintosh laryngoscopy.

After the groups completed their interventions, those who drawed envelope number 1 will be asked to intubate with Macintosh laryngoscopy using endotracheal tube introducer and those who drawed envelope number 2 will be asked to intubate with Macintosh laryngoscopy. Each doctor will be given 1 minute for each successful intervention. Each practitioner will make maximum 2 trial attempts for each method. The initiation time is considered to be taking the laryngoscopy on hand. After ventilation, the manikin's chest wall movement is considered as a successful intervention. All transactions will be recorded with a camera that is placed in the room and the participants will have the information about the presence of the camera. The first intervention success , intubation time, the number of interventions of the participants will be recorded. After the interventions are over, the participants will be asked to rate the difficulty of the ventilation methods according to the Likert scale as 1-very easy, 2-easy, 3-medium, 4-difficult 5- very difficult. In addition, they will be asked whether they have any experiences with Macintosh laryngoscopy or endotracheal tube introducer and their responses will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* novice doctors who accept to participate the study

Exclusion Criteria:

* novice doctors who won't accept to participate the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2018-03-10 (Actual); Study Completion 2018-03-10 (Actual)

PRIMARY OUTCOMES:
First pass success | 1 minute
  The primary outcome measure of the survey is determined as the first pass success of the doctors.

SECONDARY OUTCOMES:
intubation duration | 1 minute
  The initiation time is considered to be taking the laryngoscope on hand. Successful ventilation of the manikin with a balloon valve mask is considered as the ending time of the intervention.
Intervention numbers | 1 minute
  All of the interventions will be recorded with a camera
Difficulty levels of the methods | 2 minutes
  Difficulty levels of the methods on the Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Derince training and educational hospital, Kocaeli, Derince, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] Murat I, Constant I, Maud'huy H. Perioperative anaesthetic morbidity in children: a database of 24,165 anaesthetics over a 30-month period. Paediatr Anaesth. 2004 Feb;14(2):158-66. doi: 10.1111/j.1460-9592.2004.01167.x. PMID 14962332
- [Background] Bhananker SM, Ramamoorthy C, Geiduschek JM, Posner KL, Domino KB, Haberkern CM, Campos JS, Morray JP. Anesthesia-related cardiac arrest in children: update from the Pediatric Perioperative Cardiac Arrest Registry. Anesth Analg. 2007 Aug;105(2):344-50. doi: 10.1213/01.ane.0000268712.00756.dd. PMID 17646488
- [Background] Fiadjoe JE, Nishisaki A, Jagannathan N, Hunyady AI, Greenberg RS, Reynolds PI, Matuszczak ME, Rehman MA, Polaner DM, Szmuk P, Nadkarni VM, McGowan FX Jr, Litman RS, Kovatsis PG. Airway management complications in children with difficult tracheal intubation from the Pediatric Difficult Intubation (PeDI) registry: a prospective cohort analysis. Lancet Respir Med. 2016 Jan;4(1):37-48. doi: 10.1016/S2213-2600(15)00508-1. Epub 2015 Dec 17. PMID 26705976
- [Background] Jabre P, Combes X, Leroux B, Aaron E, Auger H, Margenet A, Dhonneur G. Use of gum elastic bougie for prehospital difficult intubation. Am J Emerg Med. 2005 Jul;23(4):552-5. doi: 10.1016/j.ajem.2004.12.005. PMID 16032630
- [Background] Kidd JF, Dyson A, Latto IP. Successful difficult intubation. Use of the gum elastic bougie. Anaesthesia. 1988 Jun;43(6):437-8. doi: 10.1111/j.1365-2044.1988.tb06625.x. PMID 3407866
- See also: The difficult pediatric airway - UpToDate [Internet]. Jul 31. 2017 — https://www.uptodate.com/contents/the-difficult-pediatric-airway